CLINICAL TRIAL: NCT03531476
Title: Evaluation of a Pilot Shard-care Program for Patients With Chronic Pain in the Champlain-LHIN
Acronym: Shared-Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20180238-01H
Record Dates: First submitted 2018-03-19; First posted 2018-05-21 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Chronic Pain; Quality of Life
Keywords: Mindfulness; Chronic Pain; Disability; Quality of Life; Online
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online chronic pain management program (Experimental): There is only one arm. Those who consent to participate in the study and take the online self-directed chronic pain management program with therapist support.
  Interventions: Behavioral: Online Chronic Pain Management Program

INTERVENTIONS:
Behavioral: Online Chronic Pain Management Program — With the support of a study therapist, the participant will be enrolled in a 5 week self-directed pain management program. The study therapist is a registered health professional. The program will consist of 5 weeks of mindfulness training. The mindfulness training focuses on the basics of mindfulness-based interventions including body, emotions, sensations, thoughts, compassion, pain and stress management.

SUMMARY:
The study is evaluating an intervention consisting of a five week online mindfulness program for patients being referred to the Pain Clinic and triaged to eConsult. A pain specialist will be in contact with the patient's family physician to confirm it's appropriate and then a therapist will initiate contact with the patient to assess eligibility. The therapist will be a registered health professional with experience with patients with chronic health problems and will be supporting the online program where the participant will have communication access to them. Questionnaires will be sent at three time points to assess changes.

DETAILED DESCRIPTION:
There are currently many patients waiting to be seen at The Ottawa Hospital Pain Clinic (TOHPC). However, many patients with chronic pain (CP) have exhausted medical options or could be served in the community with appropriate support for them and their family physicians (FPs). eConsult is a secure web-based platform that allows TOHPC physicians to provide pain management advice within seven days within the Champlain Local Health Integration Network (LHIN).

In order to provide enhanced care to patients and improve the uptake of eConsult for CP, the investigators have developed a shared care model for CP in the Champlain LHIN. This program combines the use of eConsult for FPs and a 5-week self-directed online CP management program with therapist support available as needed.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-years or older
* ability to understand oral and written English
* report chronic pain (≥3months)

Exclusion Criteria:

* refusal or inability to provide informed consent
* severe, unstable or untreated psychiatric conditions (ex. severe depression, psychosis, bipolar, etc.)
* does not have access to the internet or electronic device capable of watching videos

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in mean score of the Brief Pain Inventory-Interference Scale (BPI-I) | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  The interference scale measures the degree to which pain interferes in the lives of participants in 7 domains: general activity, mood, walking ability, normal work, relations with other persons, sleep and enjoyment of life on a scale from 0 to 10. The higher the score, the greater the pain interferes with patient's activities.This is a well-validated measure of pain-related disability. The minimum clinically significant difference is 1 point.

SECONDARY OUTCOMES:
Change in pain intensity, as measured by the Brief Pain Inventory. | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  The Brief Pain Inventory (BPI) Pain Severity Scale measures the severity of pain one feels at worst, at least, on average, and at the time of questionnaire completion on a scale from 0 to 10. The higher the score, the greater the pain severity.
Change in pain catastrophizing, as measured by the Pain Catastrophizing Scale | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  The Pain Catastrophizing Scale (PCS) is a 13-item instrument which will evaluate the degree to which patients have negative self-statements and catastrophizing thoughts and ideations when in pain. The PCS uses a 5-point likert scale (0=not at all, 4=all the time) and consists of three subscales (rumination, magnification, helplessness).
Change in mindfulness, as measured by the Short Form Five Facet Mindfulness Questionnaire. | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  Mindfulness will be measured using the Short Form Five Facet Mindfulness Questionnaire (FFMQ-SF). The FFMQ-SF is a 24-item instrument measuring five aspects of mindfulness: Non-reactivity to inner experience, observing, describing, acting with awareness, and non-judging of experience. Participants are asked to use a 5-point Likert-type scale (1 = never or rarely true; 5 = very often or always true) to rate how true of them they believe each statement to be.
Change in quality of life, as measured by the EuroQOL-5D | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  The EuroQOL-5D (EQ-5D) is a simple-to-use, valid, and sensitive instrument measuring quality of life. It covers 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 3 levels: no problems, some problems, or severe problems and participants use a tick box to select the statement that is most representative of their conditions. Participants are also asked to rate, using a visual analogue scale (0 to 100), their state of health.
Change from baseline in depressive symptoms, as measured by the Patient Health Questionnaire - 9 scale | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  The Patient Health Questionnaire - 9 (PHQ-9) is a 9-item scale used to assess the severity of depressive symptoms over the past two weeks and is based on Diagnostic and Statistical Manual (DSM-IV) diagnostic criteria for major depression. Total scores range from 0 to 27, and clinical cut-points correspond to mild, moderate, moderately severe, and severe depression.
Overall change in status from baseline, as measured by Patient Global Impression of Change scale | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  The participants' perceived degree of change in overall status will be measured using the Patient Global Impression of Change (PGIC) scale. The PGIC uses a 7-point likert scale (very much worse, to very much better) to measure how much the participant feels their overall status has changed since the start of the study.
Change from baseline in anxiety symptoms, as measured by the Generalized Anxiety Disorder-7 | At enrollment prior to the program, 2 weeks post-program, and at a 3-month follow-up after the program
  The Generalized Anxiety Disorder - 7 (GAD-7) is a 7-item scale used to assess the severity of anxiety symptoms over the past two weeks. Total scores range from 0 to 15, and clinical cut-points correspond to mild, moderate, and severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Poulin, PhD C. Psych, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No